CLINICAL TRIAL: NCT01617642
Title: Dental Health, Diet, Inflammation and Biomarkers in Patients With Acute Intermittent Porphyria(AIP)
Status: Active, not recruiting | Type: Observational
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2197/REK; ID/7462 SFP 1068-12 (Other Grant/Funding Number: Northern Norway Regional Health Authority)
Record Dates: First submitted 2012-06-05; First posted 2012-06-12 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Acute Intermittent Porphyria
Keywords: Porphyria; Inflammation; Diet; Iron status
MeSH Terms: conditions — Porphyria, Acute Intermittent; Porphyrias; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and plasma from 50 cases With acute intermittent porphyria and age, sex and place of 50 recidence matched controls. Urine samples. Pax tubes for RNA/DNA samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Healthy control group, matched for age and gender
- Acute intermittent porphyria: Patients with acute intermittent porphyria.

SUMMARY:
Acute intermittent porphyria (AIP) is an autosomal dominant inherited disease, which is relatively prevalent in northern Norway with a total of around 90 patients. This provides us with a special opportunity to study AIP. AIP is caused by a mutation in the porphobilinogen deaminase, an enzyme in the haem synthesis. AIP presents symptoms, particularly among fertile women and older men. Typical symptoms are abdominal pain and dark red urine, nausea, vomiting, constipation, muscle weakness and nerve damage including paraesthesia and even paresis. This is known as symptomatic or manifest AIP (MAIP). Others do not display symptoms, so-called latent AIP (LAIP). AIP attacks may be triggered by a host of medicaments which affect the haem synthesis, infections, alcohol and stress. Treatments of manifestations include high sugar intake (4 sugar lumps/hour), alternatively administer glucose and Normosang (synthetic haem arginate) by intravenous injection and removing triggering factors. Diet, glucose intake, dental health and inflammatory parameters will be examined. This study can provide new knowledge about why only some people develop symptoms of AIP. Main hypothesis: There are differences in the diet, iron status, inflammation and glucose metabolism of the MAIP group vs. the LAIP group and the control group.

DETAILED DESCRIPTION:
In a group of people with proven acute intermittent porphyria (AIP) mutation, some will remain asymptomatic, while others have repeated periods of porphyria symptoms. Glucose inhibits ALA synthetase (ALAS), the first rate-limiting enzyme in the haem synthesis. Studies of individual patients point to the fact that increased glucose and/or fructose content in the diet inhibits porphyria attacks. A high sugar intake can reduce the disease activity in patients with AIP. The diet and related biomarkers of those with latent and manifest AIP will therefore be mapped to explain why some have latent and others have manifest acute intermittent porphyria. Other studies point to the fact that people with manifest AIP who have later developed diabetes type 2 no longer have porphyria symptoms. Dental health will also be examined.

Inflammation also affects the haem synthesis. Infections and/or inflammation are known to trigger AIP attacks. The disease activity in patients with acute intermittent porphyria in relation to inflammatory status, iron status, glucose metabolism and diet will therefore be examined.

The iron metabolism is interesting to study because it is believed that the overstimulation of the haem synthesis is what triggers porphyria attacks. Haem consists of iron and protoporphyrin IX, and it is therefore possible that iron supplements in cases of iron deficiency can induce increased haem synthesis and by doing so trigger and/or aggravate AIP.

Kidney failure is a serious secondary complication in some patients with MAIP. Protein markers for kidney injury in urine will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed acute intermittent porphyria

Exclusion Criteria:

* Regulatory use of antiinflammatory drugs including steroids and NSAIDS
* Lacking consent competence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The group of patients with acute intermittent porphyria will be recruited from primary care clinics and patient organizations.
  The control group will be selected randomly from the same geographical area, matched for gender and age
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Within 2 months after inclusion
  Resting systolic and diastolic blood pressure, a number of inflammatory parameters, serum markers for iron status and inflammation
Diet registration | Within 2 months after inclusion
  Dietary registration during one week
Iron status | Within 2 months after inclusion
  Blood samples for evaluation of iron status
Inflammatory status | Within 2 months after inclusion
  Blood samples (cytokines etc) for evaluation of inflammation

SECONDARY OUTCOMES:
Dental health | Within two months after inclusion
  Evaluate dental health through clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Ole L Brekke, MD, PhD, Principal Investigator — University of Tromsø, Norway
Locations (1):
- Nordlandssykehuset HF, Bodø, Nordland, Norway

REFERENCES:
- [Background] Storjord E, Dahl JA, Landsem A, Fure H, Ludviksen JK, Goldbeck-Wood S, Karlsen BO, Berg KS, Mollnes TE, W Nielsen E, Brekke OL. Systemic inflammation in acute intermittent porphyria: a case-control study. Clin Exp Immunol. 2017 Mar;187(3):466-479. doi: 10.1111/cei.12899. Epub 2016 Dec 15. PMID 27859020
- [Background] Storjord E, Dahl JA, Landsem A, Ludviksen JK, Karlsen MB, Karlsen BO, Brekke OL. Lifestyle factors including diet and biochemical biomarkers in acute intermittent porphyria: Results from a case-control study in northern Norway. Mol Genet Metab. 2019 Nov;128(3):254-270. doi: 10.1016/j.ymgme.2018.12.006. Epub 2018 Dec 10. PMID 30583995
- [Background] Henno LT, Storjord E, Christiansen D, Bergseth G, Ludviksen JK, Fure H, Barene S, Nielsen EW, Mollnes TE, Brekke OL. Effect of the anticoagulant, storage time and temperature of blood samples on the concentrations of 27 multiplex assayed cytokines - Consequences for defining reference values in healthy humans. Cytokine. 2017 Sep;97:86-95. doi: 10.1016/j.cyto.2017.05.014. Epub 2017 Jun 6. PMID 28595117
- [Background] Storjord E, Airila-Mansson S, Karlsen K, Madsen M, Dahl JA, Landsem A, Fure H, Ludviksen JK, Fjose JO, Dickey AK, Karlsen BO, Waage Nielsen E, Mollnes TE, Brekke OL. Dental and Periodontal Health in Acute Intermittent Porphyria. Life (Basel). 2022 Aug 19;12(8):1270. doi: 10.3390/life12081270. PMID 36013449
- [Background] Storjord E, Wahlin S, Karlsen BO, Hardersen RI, Dickey AK, Ludviksen JK, Brekke OL. Potential Biomarkers for the Earlier Diagnosis of Kidney and Liver Damage in Acute Intermittent Porphyria. Life (Basel). 2023 Dec 21;14(1):19. doi: 10.3390/life14010019. PMID 38276268